CLINICAL TRIAL: NCT06617559
Title: A Prospective Comparison of Clinical and Radiological Maturation Outcomes of Autologous Quadriceps and Hamstring Tendon Grafts in Anterior Cruciate Ligament Reconstruction
Brief Title: Comparison of Autologous Quadriceps and Hamstring Tendon Grafts in Anterior Cruciate Ligament Reconstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muzaffer Agir (Other)
Collaborators: Acibadem University (Other)
Responsible Party: Sponsor-Investigator, Muzaffer Agir, Medical Doctor, Acibadem University
Organization: Acibadem University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Fulyamaslak
Record Dates: First submitted 2024-09-23; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Anterior Cruciate Ligament Injuries; Athletic Injuries; Tendon Graft; Complications
Keywords: anterior cruciate ligament reconstruction; hamstring tendons; athletic injuries
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Athletic Injuries | interventions — Anterior Cruciate Ligament Reconstruction

STUDY DESIGN:
Intervention Model Description: There are two standard autografts used for ACL reconstruction in the investigators' clinic: quadriceps and hamstring autografts. Patients will be randomly assigned to groups based on the order of their hospital admission. It is planned to have at least 25 patients in each group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- All-inside Quadriceps Tendon Graft Group (Experimental)
  Interventions: Procedure: Anterior Cruciate Ligament Reconstruction with Quadriceps Autograft
- All-inside Hamstring Tendon Graft Group (Experimental)
  Interventions: Procedure: Anterior Cruciate Ligament Reconstruction with Hamstring Autograft

INTERVENTIONS:
Procedure: Anterior Cruciate Ligament Reconstruction with Quadriceps Autograft — The investigators will perform all-inside anterior cruciate ligament reconstruction using only the tendon portion of the quadriceps tendon (without bone fragments) in this group.
  Arms: All-inside Quadriceps Tendon Graft Group
Procedure: Anterior Cruciate Ligament Reconstruction with Hamstring Autograft — The investigators will perform all-inside anterior cruciate ligament reconstruction using the hamstring tendon as a graft in this group.
  Arms: All-inside Hamstring Tendon Graft Group

SUMMARY:
With the recent technological advancements, the use of the quadriceps tendon with an all-inside technique has come to the forefront, and large-scale research has focused especially on quadriceps tendon grafts. Clinical study results have reported that the outcomes are similar to those of patellar tendon grafts and either equivalent or superior to hamstring tendon grafts.

The aim of this study is the prospective comparison of the clinical and radiological outcomes of patients who underwent anterior cruciate ligament (ACL) reconstruction with autologous hamstring and quadriceps tendon grafts.

ELIGIBILITY:
Inclusion Criteria:

* Elite athletes
* Amateur athletes
* Anterior cruciate ligament injury

Exclusion Criteria:

* Revision surgery
* Another ligament injury ( medial collateral ligament, lateral collateral ligament, etc.. )
* > Grade-2 cartilage injury
* Having previously undergone surgery on the same knee
* < 18 years age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-05-14 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Autograft Maturation | 12 months
  Comparison of different autografts maturation on MRI images. The signal-to-noise quotient formula will be used to assess graft maturation. According to the method described by Chan and Yau, the difference between the signals of the ACL graft and the quadriceps tendon will be used to evaluate maturation by relating it to the background signal.
Stability of Knee | 9 months
  Pivot shift test
Stability of Knee | 9 months
  laxity measuring with KT-1000 device
Stability of Knee | 9 months
  Lachman test

SECONDARY OUTCOMES:
Range of Motion | 6 months
  Measurement of knee flexion and extension degrees with a goniometer.
Muscle Strength | 9 months
  Measurement of quadriceps and hamstring muscle strength with Cybex test

CONTACTS AND LOCATIONS:
Locations (1):
- Acibadem Fulya Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The investigators do not plan to share de-identified individual participant data (IPD).

REFERENCES:
- [Background] Mouarbes D, Menetrey J, Marot V, Courtot L, Berard E, Cavaignac E. Anterior Cruciate Ligament Reconstruction: A Systematic Review and Meta-analysis of Outcomes for Quadriceps Tendon Autograft Versus Bone-Patellar Tendon-Bone and Hamstring-Tendon Autografts. Am J Sports Med. 2019 Dec;47(14):3531-3540. doi: 10.1177/0363546518825340. Epub 2019 Feb 21. PMID 30790526
- [Background] Lin KM, Boyle C, Marom N, Marx RG. Graft Selection in Anterior Cruciate Ligament Reconstruction. Sports Med Arthrosc Rev. 2020 Jun;28(2):41-48. doi: 10.1097/JSA.0000000000000265. PMID 32345925
- [Background] Cavaignac E, Coulin B, Tscholl P, Nik Mohd Fatmy N, Duthon V, Menetrey J. Is Quadriceps Tendon Autograft a Better Choice Than Hamstring Autograft for Anterior Cruciate Ligament Reconstruction? A Comparative Study With a Mean Follow-up of 3.6 Years. Am J Sports Med. 2017 May;45(6):1326-1332. doi: 10.1177/0363546516688665. Epub 2017 Mar 8. PMID 28273424